CLINICAL TRIAL: NCT02992912
Title: A Phase II Study to Assess the Efficacy of the Anti-PD-L1 Antibody Atezolizumab (MPDL3280A) Administered With Stereotactic Ablative Radiotherapy (SABR) in Patients With Metastatic Tumours
Brief Title: Atezolizumab With Stereotactic Ablative Radiotherapy in Patients With Metastatic Tumours
Acronym: SABR-PDL1
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-005464-42; 2335/2015 (Other: CSET number)
Record Dates: First submitted 2016-12-12; First posted 2016-12-14 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Patients With Metastatic Tumours (Colorectal Cancer, Non-small Lung Cancer, Renal Cell Carcinoma or Sarcoma )
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Renal Cell; Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1: metastatic colorectal cancer (Experimental)
  Interventions: Drug: Anti-PD-L1 antibody atezolizumab; Procedure: SABR
- Cohort 2: metastatic non-small lung cancer (Experimental)
  Interventions: Drug: Anti-PD-L1 antibody atezolizumab; Procedure: SABR
- Cohort 3: metastatic renal cell carcinoma (Experimental)
  Interventions: Drug: Anti-PD-L1 antibody atezolizumab; Procedure: SABR
- Cohort 4: metastatic sarcoma (Experimental)
  Interventions: Drug: Anti-PD-L1 antibody atezolizumab; Procedure: SABR

INTERVENTIONS:
Drug: Anti-PD-L1 antibody atezolizumab — 1200 mg every 3 weeks
Procedure: SABR — Hypofractionated SABR will be delivered at a dose of 45 Gy in 3 fractions of 15 Gy
  Other Names: Stereotactic ablative radiotherapy

SUMMARY:
Although it is usually described as an immunosuppressive modality and not thought of as immunotherapy, there are new preclinical evidences suggesting that high-dose ionizing irradiation (IR) results in direct tumour cell death and augments tumour-specific immunity, which enhances tumour control both locally and distantly. Importantly, IR effects exceed the classical cytocidal properties by also causing phenotypic changes in the fraction of surviving cells, markedly enhancing their susceptibility to T cell-mediated elimination. However, not all IR-induced modifications of the tumour and its microenvironment favor immune rejection. The tumour microenvironment is populated by various types of inhibitory immune cells including Tregs, alternatively activated macrophages, and myeloid-derived suppression cells (MDSCs), which suppress T cell activation and promote tumour outgrowth. Chiang et al. showed the accumulation of pro-tumourigenic M2 macrophages in areas of hypoxia present in irradiated tumours. IR then may also induced responses that are inadequate to maintain antitumour immunity.

Close interaction between IR, T cells, and the PD-L1/PD-1 axis exsit and provide a basis for the rational design of combination therapy with immune modulators and radiotherapy. Deng et al. demonstrate that PD-L1 was upregulated in the tumour microenvironment after IR. Moreover, administration of anti-PD-L1 enhanced the efficacy of IR through a cytotoxic T cell-dependent mechanism. Concomitant with IR-mediated tumour regression, IR and anti-PD-L1 synergistically reduced the local accumulation of tumour-infiltrating MDSCs, which suppress T cells and alter the tumour immune microenvironment. Finally, activation of cytotoxic T cells with combination therapy mediated the reduction of MDSCs in tumours through the cytotoxic actions of TNF. Sagiv-Barfi et al, also demonstrated in 5 patients receiving atezolizumab and radiation therapy, at least stabilization of systemic progression in all patients and a RECIST partial response at systemic sites in 1 patient. Transient, grade 1-2 inflammatory adverse events (fevers, flu-like symptoms) occurred with no serious immune-related toxicities. Abscopal out-field effects of irradiation has also been described in addition to a reduction in circulating MDSCs in a melanoma patient treated with the anti CTLA-4 ipilimumab and radiotherapy.

Lastly, recent evidence demonstrates that loco-regional curative treatment with stereotactic ablative radiotherapy (SABR) is a good alternative as compared with conventional 3D RT for patients with solid tumour, with durable remissions and a low toxicity profile. Many non-randomised studies have shown that SBRT for oligometastases is safe and effective, with local control rates of about 80%. Importantly, these studies also suggest that the natural history of the disease is changing, with 2-5 year progression-free survival of about 20%. For colorectal, non-small cell, and renal cell cancers, 1-year metastasis control rates ranged from 67 to 91%. Moreover, abscopal responses in the setting of immune checkpoints inhibitors and radiotherapy combinations have been made in the setting of metastatic disease event in patients with extensive tumor burden. The goal of SABR is to deliver appropriate metastasis directed radiotherapy while minimizing exposure of surrounding normal tissues. Interestingly, the dose and fractionation employed modulate RT ability to synergize with immunotherapy. Vanpouille-Box et al, showed that immune response genes were differentially expressed in irradiated tumours by 8Gyx3 but not 20Gyx1. This highlight the interest of hypofractionated SABR acting as a "in situ tumour vaccine".

As hypofractionated SABR may, in addition to its good local control, increase the effectiveness of anti PD-L1, investigators aimed to investigate the efficacy and the tolerability of the combination of anti-PD-L1 antibody with SABR.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 years of age or older.
2. Histologically or cytologically proven metastatic solid tumours including: - colorectal (CRC, Microsatellite instability negative and positive) in treatment failure as per the current standard recommendation (cohort closed to inclusions).

   * non-small cell lung cancer (NSCLC) pretreated by at least one line of treatment. Patients EGFR-mutant can be included only if they have been treated with, or developed toxicity with or refused to be treated with anti-EGFR therapy; Patients pretreated by anti-PD1, or anti-PDL1 therapeutic antibodies can be included only if they have received at least 4 months of treatment (cohort closed to inclusions).
   * renal cell carcinoma (RCC) pretreated by at least one line therapy by a tyrosin kinase inhibitor (cohort closed to inclusions).
   * metastatic sarcomas of any type (soft tissue, bone, GISTs) pretreated by at least one line of standard therapy ; at least three lines of standard TKi must be given in patients with GISTs. No enrolment restriction to certain sarcoma subtypes/groups was decided given the relative rarity of this disease type and that immunotherapy efficacy in certain histological subtypes is only preliminary (cohort closed to inclusions).
3. Patients with at least :

   * one measurable metastasis by RECIST 1.1 eligible for SABR in terms of dose constraints at organ at risk (refer to Appendix 1: Rules for SABR administration according to tumour location ; distinct criteria apply regarding lung and liver metastases) and ≤ 4 cm, and
   * one not treated measurable metastasis by RECIST 1.1. If all tumour sites are accessible to SABR, one of them will not be treated.

   Metastase located within the proximal bronchial tree as defined in RTOG 0236 (refer to Appendix 1: Rules for SABR administration according to tumour location) or within the brain are not eligible for SABR treatment in the present study. However, it can be considered as a not treated evaluable metastase.
4. WHO performance status of 0-1
5. Evaluation by a radiation oncologist within 45 days prior to study registration, including imaging workup to document metastases (cf. description in assessment section)
6. Patients must have adequate organ function defined by the following laboratory results obtained within 28 days prior to the first study treatment:

   * Absolute neutrophil count of ≥ 1500/mm3;
   * Lymphocyte count ≥ 500 mm3;
   * Platelets ≥ 100,000/mm3;
   * Hemoglobin > 9 gr/dL;
   * Clearance Creatinine ≥ 50 mL/min;
   * Total bilirubin ≤ 1.5X ULN (unless Gilbert where 3X ULN is permitted);
   * Serum ALT and AST ≤ 2.5X ULN (unless documented liver metastases where ≤ 5X ULN is permitted),
   * ALK ≤ 2.5 ULN (unless documented bone or liver metastases where ≤ 5X ULN is permitted).
7. Life expectancy of more than 3 months
8. Patients must be aware of the investigational nature of the therapy and provide written informed consent.
9. Sexually active women of childbearing potential must agree to use a highly effective method of contraception supplemented with a barrier method, or to abstain from sexual activity during the study and for at least 5 months after the last dose of atezolizumab Sexually active males patients must agree to use condom while on SABR treatment and for at least 90 days after SABR treatment. Taking into account the irradiated area, use of condom after SABR treatment can be shortened at investigator discretion. Also, their women of childbearing potential partner should use a highly effective method of contraception.

   Women who are not postmenopausal (≥ 12 months of non-therapy-induced amenorrhea) or surgically sterile must have a negative serum β-HCG pregnancy test result within 7 days prior to initiation of study drug.

   A list of highly effective birth control methods and the definition of a woman of childbearing potential are provided in the core protocol (section 4.1).
10. Patients must be free of significant comorbid conditions that would preclude safe administration or completion of protocol therapy.
11. The irradiated and unirradiated tumour sites must be accessible to tumour biopsy (additional written consent required).
12. Patients must be affiliated to a social security system

Exclusion Criteria:

1. Known allergy to anti-PD-L1 including :

   * History of severe allergic anaphylactic reactions to chimeric, human or humanized antibodies, or fusion proteins.
   * Known hypersensitivity to CHO cell products or any component of the atezolizumab formulation.
2. Pregnant or breastfeeding women
3. Any malignancy other than the disease under study in the past 5 years excepting skin cancers such as BCC or SCC.
4. Uncontrolled tumour-related pain Patients requiring pain medication must be on a stable regimen at study entry. Asymptomatic metastatic lesions whose further growth would likely cause functional deficits or intractable pain (e.g., epidural metastasis that is not presently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to enrolment.
5. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently).

   Patients with indwelling catheters (e.g., PleurX) are allowed.
6. Uncontrolled hypercalcemia (> 1.5 mmol/L ionized calcium or Ca > 12 mg/dL or corrected serum calcium > ULN) or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab.

   Patients who are receiving bisphosphonate therapy or denosumab specifically to prevent skeletal events and who do not have a history of clinically significant hypercalcemia are eligible. However, patients who are receiving denosumab prior to enrollment must be eligible to receive bisphosphonate instead and willing to switch to bisphosphonate therapy while on the study.
7. Severe, active co-morbidity, defined as follows:

   * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months prior to registration;
   * Transmural myocardial infarction within the last 6 months prior to registration;
   * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration;
   * Uncontrolled Chronic Obstructive Pulmonary Disease or other respiratory illness requiring hospitalization or precluding study therapy within 30 days prior to registration
   * History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
   * Severe hepatic disease, defined as a diagnosis of Child-Pugh Class B or C hepatic disease.
   * Known HIV positive status.
   * End-stage renal disease (i.e., on dialysis or dialysis has been recommended).
   * Patients with active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C.

   Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
8. Active or History of autoimmune or inflammatory disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with anti-phospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis (see Appendix 3 for a more comprehensive list of autoimmune diseases) Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone are eligible Patients with controlled Type 1 diabetes mellitus on a stable insulin regimen are eligible Patients with vitiligo or psoriasis or grave's disease, not requiring systemic treatment within the last 2 years, are eligible
9. Metastases located to the brain and with clinical signs and/or leptomingeal carcinomatosis, or with indistinct borders making targeting not feasible Metastases located to the brain and without clinical signs can be included.
10. Irradiation required for cord compression and for superior veina cava syndrome.
11. Irradiation by SABR should not include metastases located within 3 cm of the previously irradiated structures:

    * Spinal cord previously irradiated to > 40 Gy
    * Brachial plexus previously irradiated to > 50 Gy
    * Small intestine, large intestine, or stomach previously irradiated to > 45 Gy
    * Brainstem previously irradiated to > 50 Gy
    * Lung previously irradiated with prior V20Gy > 30%
12. Metastasis localized to the central part of the chest and requiring irradiation (see "no fly zone" in Appendix 1: Rules for SABR administration according to tumour location).
13. Any approved anticancer therapy, including chemotherapy, hormonal therapy or radiotherapy, under the following guidelines:

    * investigational or cytotoxic treatments within 4 weeks prior to the study treatment initiation and while on study treatment
    * localized palliative radiotherapy within 2 weeks prior to the study treatment initiation and while on study treatment
    * any approved TKIs within 3 weeks prior to the study treatment initiation and while on study treatment however Hormone-replacement therapy or oral contraceptives are allowed
14. Administration of a live, attenuated vaccine within 4 weeks prior to Cycle 1, Day 1 or anticipation that such a live attenuated vaccine will be required during the study.
15. Influenza vaccination should be given during influenza season only (example: approximately October to March in the Northern Hemisphere). Patients must not receive live, attenuated influenza vaccine (e.g., FluMist®) within 4 weeks prior to Cycle 1, Day 1 or at any time during the study
16. Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumour necrosis factor [TNF] agents) within 2 weeks prior to Cycle 1, Day 1, or anticipated requirement for systemic immunosuppressive medications during the trial Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled in the study The use of inhaled corticosteroids for chronic obstructive pulmonary disease, mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension, and low-dose supplemental corticosteroids for adrenocortical insufficiency are allowed.
17. Patient already enrolled in another therapeutic trial involving an investigational substance, and when such a substance has been taken during the previous 4 weeks.
18. Persons deprived of their freedom or under guardianship, or for whom it would be impossible to undergo the medical follow-up required by the trial, for geographic, social or psychological reasons
19. Prior treatment with CD137 agonists or immune checkpoint blockade therapies, anti-PD1, or anti-PDL1 therapeutic antibodies Only patients with non-small cell lung cancer are allowed to have received anti-PD1, or anti-PDL1 therapeutic antibodies. Subjects who have received prior anti-PD-1/L1 therapies must have received at least 4 months of treatment.

    Patients who have received prior treatment with anti-CTLA-4 may be enrolled, provided at least 5 half-lives (approximately 75 days) have elapsed from the last dose of anti-CTLA-4 to the first dose of atezolizumab and there was no history of severe immune-mediated adverse effects from anti-CTLA-4 (NCI CTCAE Grade 3 and 4)
20. Treatment with systemic immunostimulatory agents (including but not limited to interferon-alpha (IFN-α) and interleukin-2 (IL-2) within 4 weeks or five half-lives of the drug (whichever is shorter) prior to Cycle 1, Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 1 year after inclusion
  Using RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France

REFERENCES:
- [Derived] Levy A, Morel D, Texier M, Rodriguez-Ruiz ME, Bouarroudj L, Bouquet F, Bustillos A, Quevrin C, Clemenson C, Mondini M, Meziani L, Sun R, Zaghdoud N, Tselikas L, Assi T, Faron M, Honore C, Ngo C, Verret B, Le Pechoux C, Le Cesne A, Ginhoux F, Massard C, Bahleda R, Deutsch E. Monocyte-lineage tumor infiltration predicts immunoradiotherapy response in advanced pretreated soft-tissue sarcoma: phase 2 trial results. Signal Transduct Target Ther. 2025 Mar 17;10(1):103. doi: 10.1038/s41392-025-02173-3. PMID 40097400
- [Derived] Levy A, Morel D, Texier M, Sun R, Durand-Labrunie J, Rodriguez-Ruiz ME, Racadot S, Supiot S, Magne N, Cyrille S, Louvel G, Massard C, Verlingue L, Bouquet F, Bustillos A, Bouarroudj L, Quevrin C, Clemenson C, Mondini M, Meziani L, Tselikas L, Bahleda R, Hollebecque A, Deutsch E. An international phase II trial and immune profiling of SBRT and atezolizumab in advanced pretreated colorectal cancer. Mol Cancer. 2024 Mar 23;23(1):61. doi: 10.1186/s12943-024-01970-8. PMID 38519913